CLINICAL TRIAL: NCT01519310
Title: Gut Flora Dependent Metabolism of Dietary Phosphatidylcholine and Cardiovascular Disease
Acronym: Glory
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-988
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Nutrition
Keywords: choline metabolism; gut flora; phosphatidylcholine; lecithin
MeSH Terms: interventions — Anti-Bacterial Agents; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): Group 1 (Antibiotics/probioitic):
  Interventions: Other: Antibiotic (metronidazole and ciprofloxacin)/probiotic
- Group 2 (Active Comparator): Group 2 (Antibiotics/no-probiotic):
  Interventions: Other: Antibiotic (metronidazole and ciprofloxacin)/probiotic
- Group 3 (Active Comparator): Group 3 (no-Antibiotics/probiotic):
  Interventions: Other: Antibiotic (metronidazole and ciprofloxacin)/probiotic

INTERVENTIONS:
Other: Antibiotic (metronidazole and ciprofloxacin)/probiotic — Antibiotic cocktail/yogurt as follows:
  Group 1: antibiotics for 1 week, followed by probiotics for 3 weeks; Group 2: antibiotics for 1 week, followed by no probiotics for 3 weeks. Group 3: no antibiotics for 1 week, followed by probiotics for 3 weeks.

SUMMARY:
The purpose of this study is to see if intestinal bacteria plays a role in choline metabolism (a form of choline monitored in this study is called phosphatidylcholine, also known as lecithin). This study will help to determine if choline metabolism is affected by short-term antibiotic therapy, and/or can be altered by probiotic therapy (e.g. in the form of eating yogurt).

DETAILED DESCRIPTION:
The purpose of this study is to see if intestinal bacteria plays a role in choline metabolism (a form of choline monitored in this study is called phosphatidylcholine, also known as lecithin). This study will help to determine if choline metabolism is affected by short-term antibiotic therapy, and/or can be altered by probiotic therapy (e.g. in the form of eating yogurt).

Metabolism is a process that turns foods we eat into fuel for our bodies. Choline is nutrient found in a type of fat commonly found in foods. There is evidence that choline metabolism by bacteria in the intestines may be linked to cardiac risk.

The purpose of this study is to see if intestinal bacteria plays a role in choline metabolism (a form of choline monitored in this study is called phosphatidylcholine, also known as lecithin). This study will help to determine if choline metabolism is affected by short-term antibiotic therapy, and/or can be altered by probiotic therapy (e.g. in the form of eating yogurt).

This single center study will randomize 30 normal, healthy volunteers to 1 of 3 groups:

Group 1: antibiotics for 1 week, followed by probiotics for 3 weeks; Group 2: antibiotics for 1 week, followed by no probiotics for 3 weeks. Group 3: no antibiotics for 1 week, followed by probiotics for 3 weeks.

The antibiotics to be used will be metronidazole (500 mg twice daily) and ciprofloxacin (500 mg daily) for one week. The probiotics to be used will be one serving size of standard flavored yogurt (approximately 170 g) twice daily for up to three weeks.

Study visits will occur at baseline, 1 week, and 4 weeks. Blood and urine samples will be collected at the start of each visit. Subjects will then eat 2 hard boiled eggs and be given a standard medical isotope. Additional blood samples will be obtained at 1, 2, 3, 4, and 6 hours, and a urine sample will be collected at 6 hours. Samples will be analyzed for choline levels, its byproducts, and isotope levels.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or above.
* Able to provide informed consent and comply with study protocol

Exclusion Criteria:

* Significant chronic illness or end-organ dysfunction, including known history of heart failure, renal failure, pulmonary disease, or hematologic diseases.
* Active infection or received antibiotics within 2 months of study enrollment
* Use of OTC probiotic within past 2 months, or ingestion of yogurt within past month
* Chronic gastrointestinal disorders, or intolerance to probiotic therapy
* Allergies to eggs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Primary Outcome | December 2016
  Phosphatidylcholine derived gut flora metabolites

SECONDARY OUTCOMES:
Secondary Outcome Measures | December 2016
  Cardiometabolic risk markers

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States